CLINICAL TRIAL: NCT02043600
Title: Randomized-controlled Trial of Yoga for Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Deutsche Morbus Crohn / Colitis ulcerosa Vereinigung DCCV (Unknown)
Responsible Party: Principal Investigator, Holger Cramer, Postdoctoral Researcher, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-5560-BO
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Colitis, Ulcerative
Keywords: Colitis, ulcerative; Yoga
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Yoga; Self Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental)
  Interventions: Behavioral: Yoga
- Self-care (Active Comparator)
  Interventions: Behavioral: Self-care

INTERVENTIONS:
Behavioral: Yoga — 12-week Hatha Yoga intervention 90 minutes once a week
  Arms: Yoga
Behavioral: Self-care — Self-care books are provided for self-directed use
  Other Names: Self-care book
  Arms: Self-care

SUMMARY:
The aim of this randomized trial is to investigate the effects of a 12-week yoga intervention compared to self-care on quality of life, stress, psychological health, and physiological parameters in 77 patients with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis (clinical, endoscopic and histological diagnosis)
* Disease duration at least 12 months
* Clinical remission for at least 4 weeks and less than 12 months
* CAI < 5
* IBDQ < 170
* Physical and mental ability to perform yoga
* No regular practice of yoga or Pilates in the previous 12 months

Exclusion Criteria:

* Clinically active disease (CAI > 4 Rachmilewitz)
* Complete resection of the colon
* Acute, infectious or chronic active ulcerative colitis
* Severe disease precluding yoga practice
* Malignancy with a disease-free survival < 5 years except curatively treated basalioma of the skin
* Alcohol or drug abuse
* Dementia
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-02; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Disease-specific quality of life | 3 months
  Inflammatory Bowel Disease Questionnaire (IBDQ)

SECONDARY OUTCOMES:
Disease-specific quality of life | 6 months
  Inflammatory Bowel Disease Questionnaire (IBDQ)
Generic quality of life | 3 months
  36-Item Short Form Health Survey (SF-36)
Generic quality of life | 6 months
  36-Item Short Form Health Survey (SF-36)
Anxiety/depression | 3 months
  Hospital Anxiety and Depresion Scale (HADS)
Anxiety/depression | 6 months
  Hospital Anxiety and Depresion Scale (HADS)
Subjective stress | 3 months
  Perceived Stress Scale (PSS)
Subjective stress | 6 months
  Perceived Stress Scale (PSS)
Subjective stress | 3 months
  Perceived Stress Questionnaire (PSQ)
Subjective stress | 6 months
  Perceived Stress Questionnaire (PSQ)
Positive/negative affect | 3 months
  Positive and Negative Affect Schedule (PANAS)
Positive/negative affect | 6 months
  Positive and Negative Affect Schedule (PANAS)
Body awareness | 3 months
  Body Awareness Questionnaire (BAQ)
Body awareness | 6 months
  Body Awareness Questionnaire (BAQ)
Body responsiveness | 3 months
  Body Responsiveness Scale (BRS)
Body responsiveness | 6 months
  Body Responsiveness Scale (BRS)
Self-efficacy | 3 months
  General Self-Efficacy Scale
Self-efficacy | 6 months
  General Self-Efficacy Scale
C-reactive protein | 3 months
  C-reactive protein
C-reactive protein | 6 months
  C-reactive protein
Blood sedimentation rate | 3 months
  Blood sedimentation rate
Blood sedimentation rate | 6 months
  Blood sedimentation rate
Faecal calprotectin | 3 months
  Faecal calprotectin
Faecal calprotectin | 6 months
  Faecal calprotectin
Faecal lactoferrin | 3 months
  Faecal lactoferrin
Faecal lactoferrin | 6 months
  Faecal lactoferrin
Faecel PMN-elastase | 3 months
  Faecel PMN-elastase
Faecel PMN-elastase | 6 months
  Faecel PMN-elastase
Disease activity | 3 months
  Clinical Activity Index (CAI-Rachmilewitz)
Disease activity | 6 months
  Clinical Activity Index (CAI-Rachmilewitz)
Salivary cortisol level | 3 months
  Salivary cortisol level - cortisol awakening response
Steroid sensitivity | 3 months
  Steroid sensitivity (IC50)
Andrenergic sensitivity | 3 months
  Andrenergic sensitivity (IC50)
Cholinergic sensitivity | 3 months
  Cholinergic sensitivity (IC50)
Safety | 3 months
  Number of patients with adverse events/serious adverse events
Safety | 6 months
  Number of patients with adverse events/serious adverse events
Hemogram | 3 months
  Hemogram
Hemogram | 6 months
  Hemogram

OTHER OUTCOMES:
Adherence | 3 months
  Intervention adherence (number of sessions attended and home practice diary)

CONTACTS AND LOCATIONS:
Overall Officials: Holger Cramer, PhD, Principal Investigator — Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen, Essen, Germany; Jost Langhorst, MD, Study Director — Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen, Essen, Germany
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen, Essen, Germany

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Koch AK, Schols M, Langhorst J, Dobos G, Cramer H. Perceived stress mediates the effect of yoga on quality of life and disease activity in ulcerative colitis. Secondary analysis of a randomized controlled trial. J Psychosom Res. 2020 Mar;130:109917. doi: 10.1016/j.jpsychores.2019.109917. Epub 2019 Dec 31. PMID 31927346
- [Derived] Cramer H, Schafer M, Schols M, Kocke J, Elsenbruch S, Lauche R, Engler H, Dobos G, Langhorst J. Randomised clinical trial: yoga vs written self-care advice for ulcerative colitis. Aliment Pharmacol Ther. 2017 Jun;45(11):1379-1389. doi: 10.1111/apt.14062. Epub 2017 Apr 5. PMID 28378342